CLINICAL TRIAL: NCT00617201
Title: Evaluation of Atomoxetine for Cocaine Dependence: A Pilot Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sharon Walsh (Other)
Collaborators: Eli Lilly and Company (Industry); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Sharon Walsh, Director Center on Drug and Alcohol Research, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: #07-0041; R01DA022191 (NIH)
Record Dates: First submitted 2008-02-05; First posted 2008-02-15 (Estimated); Results first posted 2012-12-11 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Substance Abuse
Keywords: cocaine; dependence; stimulants
MeSH Terms: conditions — Substance-Related Disorders | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Atomoxetine
  Interventions: Drug: atomoxetine
- 2 (Placebo Comparator): Matched Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: atomoxetine — Once daily oral dosing
  Other Names: Straterra
  Arms: 1
Drug: placebo — Once daily oral dosing - matched placebo
  Arms: 2

SUMMARY:
This placebo-controlled, double-blind, randomized pilot clinical trial will evaluate atomoxetine (Strattera®) for the treatment of cocaine dependence. Cocaine-dependent individuals, who are healthy and are seeking treatment for their substance abuse, will be randomized to receive either atomoxetine (n=25) or a matched-placebo (n=25) during a trial lasting 12 weeks; there will be a double-blind, ascending dose lead-in order to achieve maintenance on the assigned active dose safely. Contingency management procedures will be used to reinforce attendance and compliance with study procedures. Primary outcome measures will include urinalysis data assessing cocaine use.

ELIGIBILITY:
Inclusion Criteria:

* Seeking treatment for cocaine dependence
* Must have used cocaine in the past 30 days

Exclusion Criteria:

* Physical dependence on any drug requiring medical management
* Any major medical or psychiatric disorder that would be contraindicated for participation
* Cardiovascular disease
* Seizures or significant head injuries
* Currently taking atomoxetine
* Pregnant or breast-feeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2007-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon L Walsh, Ph.D., Principal Investigator — University of Kentucky
Locations (1):
- Straus Research Building, Lexington, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult volunteers ages 18-60 reporting cocaine use in the preceding 30 days who met the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-IV) criteria for and were seeking treatment for cocaine dependence were recruited through advertisements and word-of-mouth to a research clinic.
Pre-assignment Details: Exclusions included dependence on any drug requiring detoxification, other Axis I disorders, medical problems, pregnant or lactating females, Cytochrome P450 2D6 inhibitors/inducers, monoamine oxidase inhibitors or selective serotonin reuptake inhibitors. Enrollment in other drug treatment programs urine samples required for parole/probation.
Groups:
- Atomoxetine (80 mg/Day): Active drug
  atomoxetine : Once daily oral dosing
- Matched Placebo: Matched Placebo
  placebo : Once daily oral dosing - matched placebo
Period: Overall Study
Arm/Group | Atomoxetine (80 mg/Day) | Matched Placebo
Started | 25 | 25
Completed | 16 | 12
Not Completed | 9 | 13
Not completed — Lost to Follow-up | 9 | 13

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Matched placebo
- Atomoxetine: Atomoxetine (80 mg/day)
- Total: Total of all reporting groups
Arm/Group | Placebo | Atomoxetine | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (1.6) | 44.5 (1.6) | 42 (1.7)
Sex/Gender, Customized [Number; unit: participants]
  Female | 8 | 19 | 27
  Male | 17 | 6 | 23
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: % Urine Samples Negative for Cocaine
Description: Total % urine samples negative for benzoylecgonine over the 12-week trial
Time Frame: Urines were collected 3 times per week (e.g., Monday, Wednesday and Friday) for 12 weeks
Population: Intent-to-treat analysis included all subjects with missing urine sample counted as positive.
Measure: Number; unit: percentage of positive urine samples
Units Other Than Participants: Urine samples
Groups:
- Atomoxetine: 80 mg/day (after intial 4-day run up)
Arm/Group | Placebo | Atomoxetine
Number analyzed (Participants) | 25 | 25
Number analyzed (Urine samples) | 598 | 537
percentage of positive urine samples | .67 | .74

2. Secondary Outcome: Retention
Description: Trial retention- those who complete the 12 week dosing period
Time Frame: 12-weeks
Population: those completing the 12-week study after randomization
Measure: Mean (Standard Error); unit: days
Arm/Group | Placebo | Atomoxetine
Number analyzed (Participants) | 25 | 25
days | 57.4 (7) | 51.6 (6.7)

ADVERSE EVENTS:
Arm/Group | Atomoxetine (80 mg/Day) | Matched Placebo
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No